CLINICAL TRIAL: NCT05186818
Title: A Phase 3, Multi-Center, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of CK-3773274 in Adults With Symptomatic Hypertrophic Cardiomyopathy and Left Ventricular Outflow Tract Obstruction
Brief Title: Aficamten vs Placebo in Adults With Symptomatic Obstructive Hypertrophic Cardiomyopathy (SEQUOIA-HCM)
Acronym: SEQUOIA-HCM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Collaborators: Corxel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CY 6031; 2021-003536-92 (EudraCT Number)
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy (oHCM)
Keywords: Obstructive Hypertrophic Cardiomyopathy; oHCM; CK-3773274; CK-274; Aficamten; SEQUOIA-HCM; CY 6031; SEQUOIA
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aficamten up to 20 mg (Experimental): Participants received 5 mg, 10 mg, 15 mg, or 20 mg of aficamten; dose levels were guided by echocardiography assessments. Treatment was administered for up to 24 weeks.
  Interventions: Drug: Aficamten (5 mg, 10 mg, 15 mg, and 20 mg)
- Placebo to match aficamten (Placebo Comparator): Participants received placebo for up to 24 weeks.
  Interventions: Drug: Placebo to match aficamten

INTERVENTIONS:
Drug: Aficamten (5 mg, 10 mg, 15 mg, and 20 mg) — Aficamten tablets were administered orally once daily.
  Other Names: CK-3773274
  Arms: Aficamten up to 20 mg
Drug: Placebo to match aficamten — Placebo tablets were administered orally once daily.
  Other Names: Placebo
  Arms: Placebo to match aficamten

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of aficamten (CK-3773274) versus placebo in adults with symptomatic hypertrophic cardiomyopathy (HCM) and left ventricular outflow tract obstruction.

DETAILED DESCRIPTION:
CY 6031 was a Phase 3, randomized, placebo-controlled, double-blind, multi-center trial in participants with symptomatic oHCM. Eligible participants were randomized in a 1:1 ratio to receive aficamten or placebo. Randomization was stratified by use of beta-blockers (yes or no) and cardiopulmonary exercise testing (CPET) exercise modality (treadmill or bicycle). Enrollment limits were applied as follows: participants taking beta-blockers were capped at approximately 70% of total enrollment; participants taking disopyramide were capped at approximately 10% of total enrollment; participants with persistent atrial fibrillation (AF) at screening were capped at approximately 15% of total enrollment; and participants using the bicycle CPET exercise modality were capped at approximately 50% of total enrollment.

Investigational product (IP) was administered orally once daily (QD) with or without food for 24 weeks. During the initial 6 weeks of the treatment period, IP doses were individually titrated at Weeks 2, 4, and 6 based on echocardiography-guided criteria. Dose escalation at Weeks 2, 4, and 6 occurred only if a participant had a Valsalva LVOT-G ≥ 30 mmHg and a biplane left ventricular ejection fraction (LVEF) ≥ 55%. Echocardiograms were performed at each subsequent visit during the trial, and the IP dose was down-titrated if the LVEF was < 50%. The primary endpoint of peak oxygen uptake (pVO2) was measured by CPET at screening and at the end of treatment (Week 24). A participant's background HCM therapy was individually optimized according to local practice prior to enrollment in the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females between 18 and 85 years of age, inclusive, at screening.
* Body mass index <35 kg/m2.
* Diagnosed with HCM per the following criteria:

  * Has LV hypertrophy and non-dilated LV chamber in the absence of other cardiac disease and
  * Has an end-diastolic LV wall thickness as measured by the echocardiography core laboratory of:

    * ≥15 mm in one or more myocardial segments OR
    * ≥13 mm in one or more wall segments and a known-disease-causing gene mutation or positive family history of HCM
* Has resting LVOT-G ≥30 mmHg and post-Valsalva LVOT G ≥50 mmHg during screening as determined by the echocardiography core laboratory.
* LVEF ≥60% at screening as determined by the echocardiography core laboratory.
* NYHA Functional Class II or III at screening.
* Hemoglobin ≥10g/dL at screening.
* Respiratory exchange ratio (RER) ≥1.05 and pVO2 ≤90% predicted on the screening CPET per the core laboratory.
* Patients on beta-blockers, verapamil, diltiazem, or disopyramide should have been on stable doses for >6 weeks prior to randomization and anticipate remaining on the same medication regimen during the trial. Patients treated with disopyramide must also be concomitantly treated with a beta blocker and/or calcium channel blocker.

Key Exclusion Criteria:

* Known or suspected infiltrative, genetic or storage disorder causing cardiac hypertrophy that mimics oHCM (eg, Noonan syndrome, Fabry disease, amyloidosis).
* Significant valvular heart disease (per investigator judgment).

  * Moderate-severe valvular aortic stenosis.
  * Moderate-severe mitral regurgitation not due to systolic anterior motion of the mitral valve.
* History of LV systolic dysfunction (LVEF <45%) or stress cardiomyopathy at any time during their clinical course.
* Inability to exercise on a treadmill or bicycle (eg, orthopedic limitations).
* Has been treated with septal reduction therapy (surgical myectomy or percutaneous alcohol septal ablation) or has plans for either treatment during the trial period.
* Documented paroxysmal atrial fibrillation during the screening period.
* Paroxysmal or permanent atrial fibrillation is only excluded IF:

  * rhythm restoring treatment (eg, direct-current cardioversion, atrial fibrillation ablation procedure, or antiarrhythmic therapy) has been required ≤6 months prior to screening.
  * rate control and anticoagulation have not been achieved for at least 6 months prior to screening.
* History of syncope or sustained ventricular tachyarrhythmia with exercise within 6 months prior to screening.
* Has received prior treatment with CK-3773274 or mavacamten.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen uptake (pVO2) by cardiopulmonary exercise testing (CPET) | Baseline to Week 24
  Effect of CK-3773274 on exercise capacity in patients with symptomatic oHCM

SECONDARY OUTCOMES:
Change in Kansas City Cardiomyopathy Questionnaire - Clinical Summary Score (KCCQ-CSS) | Baseline to Week 12 and Week 24
  Effect of CK-3773274 on patient health status
Proportion of patients with ≥1 class improvement in New York Heart Association (NYHA) Functional Class | Baseline to Week 12 and Week 24
  Effect of CK-3773274 on NYHA Functional Classification
Change in post-Valsalva left ventricular outflow tract gradients (LVOT-G) | Baseline to Week 12 and Week 24
  Effect of CK-3773274 on post-Valsalva LVOT-G
Proportion of patients with post-Valsalva LVOT G <30 mmHg | Baseline to Week 12 and Week 24
  Effect of CK-3773274 on post-Valsalva LVOT-G
Change in total workload during CPET | Baseline to Week 24
  Effect of CK-3773274 on exercise capacity
Duration of eligibility for septal reduction therapy (SRT) | Baseline to Week 24
  Effect of CK-3773274 on duration of eligibility for septal reduction therapy

CONTACTS AND LOCATIONS:
Overall Officials: Cytokinetics MD, Study Director — Cytokinetics
Locations (113):
- United States (48):
  - Alaska Heart and Vascular Institute, Anchorage, Alaska
  - UC San Diego Health - Sulpizio Cardiovascular Center, La Jolla, California
  - Cedars-Sinai Medical Center - Smidt Heart Institute Clinic, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Stanford University Hospital, Stanford, California
  - Yale School of Medicine, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Holy Cross Hospital / Cardiology Associates, Fort Lauderdale, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Emory Clinic, Atlanta, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - MedStar Medical Group Cardiology at Union Memorial, Baltimore, Maryland
  - Medstar Franklin Square Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - Spectrum Health Medical Group Cardiovascular Medicine, Grand Rapids, Michigan
  - M Health Fairview University of Minnesota Medical Center - East Bank, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - NYU Langone Health, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center/NY Presbyterian Hospital, New York, New York
  - Westchester Medical Center, Valhalla, New York
  - Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - Sanger Heart and Vascular Institute - HCM Clinic, Charlotte, North Carolina
  - Duke Health Center Arringdon, Morrisville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Ascension St. John Clinical Research Institute, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania (University of Pennsylvania School of Medicine), Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Stern Cardiovascular Foundation, Inc, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - University of Virginia Health System University Hospital, Charlottesville, Virginia
  - University of Washington Medical, Seattle, Washington
  - Froedtert Hospital, Milwaukee, Wisconsin
- China (9):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Nanfang Hospital Southern Medical University, Guanzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital of the Central South University, Changsha, Hunan
  - The First Hospital of Jinlin University, Changchun, Jinlin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
- Czechia (2):
  - Charles University, Prague
  - Interni klinika kardiologie a angiologie, Prague
- Denmark (4):
  - Aalborg University Hospital, Department of Cardiology, Aalborg
  - Department of Cardiology Aarhus University Hospital, Aarhus
  - Hjertecentret (The Heart Center), Copenhagen
  - Copenhagen University Hospital, Copenhagen
- France (8):
  - Hopital Universitaire de Rangueil (CHU de Toulouse) Service de Cardiologie, Toulouse, Cedex
  - CHU de Marseille - Hopital de la Timone Service de cardiologie, Marseille
  - CHU de Nantes, Nantes
  - Hopital Lariboisiere, Service de Cardiologie, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - CHU Pitie-Salpetriere, Centre de reference maladies cardiaques hereditaires ou rares, Paris
  - CHU de Bordeaux Hopital Cardiologique Haut-Leveque, Pessac
  - CHU du Haut Lveque Cardiologie, Pessac
- Germany (9):
  - Kerckhoff-Klinik GmbH Abteilung Administration Forschung und Lehre, Bad Nauheim
  - Charite-Universitaetsmedizin Berlin Campus Virchow-Klinikum (CVK) Medizinische Klinik mit Schwerpunkt Kardiologie, Berlin
  - Universitaetsklinikum Essen Westdeutsches Herz-Gefaesszentrum, Essen
  - Klinikumder Georg-August-Universitaet, Göttingen
  - Universitaetsmedizin Goettingen, Göttingen
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Jena Klinik fuer Innere Medizin 1, Jena
  - Unniversitaetsklinikum Magdeburg Klinik fur Kardiologie und Anglologie, Magdeburg
  - Universitätsklinikum Würzburg, Würzburg
- Semmelweis Egyetem Varosmajori Sziv es Ergyogyasazati Klinika, Budapest, Hungary
- Israel (5):
  - The Olga & Lev Leviev Heart Center The Chaim Sheba Medical Center, Ramat Gan, Tel Hasomer
  - The Barzilai University Medical Center, Ashkelon
  - Hadassah Medical Center- Ein Kerem, Jerusalem
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
- Italy (4):
  - UOC Cardiologica Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero Universitaria Careggi Dipartimento Cardiotoracovascolare - Cardiomiopatie Unit, Florence
  - Fondazione toscana Gabriele Monesterio per la ricarca medica Dipartimento Cardiotoracico UOC Cardiologia e Medicina Cardiovasculare Ospedale San Cataldo, Pisa
  - Dipartimento di Medicina Clinica e Molecolare Universita Sapienza di Roma Unita di Terapia Intensiva Cardiologica Azienda Ospedaliero Universitaria Sant'Andrea, Roma
- Netherlands (3):
  - Amsterdam UMC, location AMC, Amsterdam
  - University Hospital Maastricht, Maastricht
  - Erasmus Medical Center, Rotterdam
- Poland (3):
  - Narodowy Instytut Kardiologii Stefana Kardynała Wyszynskiego- Panstwowy Instytut Badawczy, Warsaw, Masovian Voivodeship
  - Kardio Brynow S.C, Katowice
  - Krakowskie Centrum, Krakow
- Portugal (2):
  - Centro Hospitalar Do Baixo Vouga, EPE AV ARTUR RAVARA, Aveiro
  - Hospital da Luz, Lisbon
- Spain (7):
  - Complejo Hospitalario Universitario, A Coruña, La Coruna
  - Hospital Universitario Puerta de Hierro, Madrid, Majadahonda
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clinico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Universitario Son Llatzer Secretaria de Cardiologia, Palma
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena-merge, Seville
- United Kingdom (8):
  - Queen Elizabeth Hospital Birmingham University Hospitals Birmingham NHS Foundation Trust, Edgbaston, Birmingham
  - Queen Elizabeth University Hospital - HWS Greater Glasgow and Clyde, Glasgow
  - Liverpool Heart and Chest Hospital - Liverpool Heart and Chest Hospital NHS Foundation Trust- HWS Greater Glasgow and Clyde, Liverpool
  - Barts Health NS Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Royal Brompton Hospital, London
  - Oxford Centre for Clinical Magnetic Resonance Research, Oxford
  - Radcliffe Department of Medicine, Oxford

REFERENCES:
- [Derived] Kaski JP, Kantor PF, Nakano SJ, Olivotto I, Russell MW, Godown J, Chiu M, German P, Heitner SB, Jacoby DL, Kupfer S, Lutz J, Maharao N, Malik FI, Melloni C, Nieto Morales PF, Simkins T, Wei J, Ho CY; CEDAR-HCM Investigators. Efficacy and Safety of Aficamten in Children and Adolescents With Obstructive Hypertrophic Cardiomyopathy: Study Design and Rationale of CEDAR-HCM. Circ Heart Fail. 2025 Dec 5:e013418. doi: 10.1161/CIRCHEARTFAILURE.125.013418. Online ahead of print. PMID 41347307
- [Derived] Campain J, Griskowitz C, Newlands C, Claggett BL, Kulac IJ, McGinnis S, Giverts I, Moreno F, Minasian A, Prasad C, Rupert L, Landsteiner I, Iskenderian N, Coats CJ, Lee MMY, Maron MS, Owens AT, Jacoby DL, Heitner SB, Kupfer S, Malik FI, Wohltman A, Malhotra R, Lewis GD. Characterization and Application of Novel Exercise Recovery Patterns That Reflect Cardiac Performance: A Substudy of the SEQUOIA-HCM Trial. Circulation. 2025 Oct 7;152(14):990-1002. doi: 10.1161/CIRCULATIONAHA.124.073585. Epub 2025 Sep 5. PMID 40910168
- [Derived] Maron MS, Masri A, Nassif ME, Barriales-Villa R, Abraham TP, Arad M, Cardim N, Choudhury L, Claggett B, Coats CJ, Dungen HD, Garcia-Pavia P, Hagege AA, Januzzi JL, Kulac I, Lee MMY, Lewis GD, Ma CS, Michels M, Oreziak A, Owens AT, Spertus JA, Solomon SD, Tfelt-Hansen J, van Sinttruije M, Veselka J, Watkins HC, Jacoby DL, Heitner SB, Kupfer S, Malik FI, Meng L, Wohltman A, Olivotto I; SEQUOIA-HCM Investigators. Impact of Aficamten on Disease and Symptom Burden in Obstructive Hypertrophic Cardiomyopathy: Results From SEQUOIA-HCM. J Am Coll Cardiol. 2024 Nov 5;84(19):1821-1831. doi: 10.1016/j.jacc.2024.09.003. Epub 2024 Sep 30. PMID 39352339
- [Derived] Lee MMY, Masri A, Nassif ME, Barriales-Villa R, Abraham TP, Claggett BL, Coats CJ, Gimeno JR, Kulac IJ, Landsteiner I, Ma C, Maron MS, Olivotto I, Owens AT, Solomon SD, Veselka J, Jacoby DL, Heitner SB, Kupfer S, Malik FI, Meng L, Wohltman A, Lewis GD; SEQUOIA-HCM Investigators. Aficamten and Cardiopulmonary Exercise Test Performance: A Substudy of the SEQUOIA-HCM Randomized Clinical Trial. JAMA Cardiol. 2024 Nov 1;9(11):990-1000. doi: 10.1001/jamacardio.2024.2781. PMID 39230885
- [Derived] Sherrod CF 4th, Saberi S, Nassif ME, Claggett BL, Coats CJ, Garcia-Pavia P, Januzzi JL, Lewis GD, Ma C, Maron MS, Miao ZM, Olivotto I, Veselka J, Butzner M, Jacoby DL, Heitner SB, Kupfer S, Malik FI, Meng L, Wohltman A, Spertus JA. Effect of Aficamten on Health Status Outcomes in Obstructive Hypertrophic Cardiomyopathy: Results From SEQUOIA-HCM. J Am Coll Cardiol. 2024 Nov 5;84(19):1773-1785. doi: 10.1016/j.jacc.2024.08.014. Epub 2024 Sep 1. PMID 39217569
- [Derived] Masri A, Cardoso RN, Abraham TP, Claggett BL, Coats CJ, Hegde SM, Kulac IJ, Lee MMY, Maron MS, Merkely B, Michels M, Olivotto I, Oreziak A, Jacoby DL, Heitner SB, Kupfer S, Malik FI, Meng L, Solomon SD, Wohltman A, Kwong RY, Kramer CM; SEQUOIA-HCM Investigators. Effect of Aficamten on Cardiac Structure and Function in Obstructive Hypertrophic Cardiomyopathy: SEQUOIA-HCM CMR Substudy. J Am Coll Cardiol. 2024 Nov 5;84(19):1806-1817. doi: 10.1016/j.jacc.2024.08.015. Epub 2024 Sep 1. PMID 39217563
- [Derived] Hegde SM, Claggett BL, Wang X, Jering K, Prasad N, Roshanali F, Masri A, Nassif ME, Barriales-Villa R, Abraham TP, Cardim N, Coats CJ, Kramer CM, Maron MS, Michels M, Olivotto I, Saberi S, Jacoby DL, Heitner SB, Kupfer S, Meng L, Wohltman A, Malik FI, Solomon SD; SEQUOIA-HCM Investigators. Impact of Aficamten on Echocardiographic Cardiac Structure and Function in Symptomatic Obstructive Hypertrophic Cardiomyopathy. J Am Coll Cardiol. 2024 Nov 5;84(19):1789-1802. doi: 10.1016/j.jacc.2024.08.002. Epub 2024 Sep 1. PMID 39217556
- [Derived] Coats CJ, Masri A, Nassif ME, Barriales-Villa R, Arad M, Cardim N, Choudhury L, Claggett B, Dungen HD, Garcia-Pavia P, Hagege AA, Januzzi JL, Lee MMY, Lewis GD, Ma CS, Maron MS, Miao ZM, Michels M, Olivotto I, Oreziak A, Owens AT, Spertus JA, Solomon SD, Tfelt-Hansen J, van Sinttruije M, Veselka J, Watkins H, Jacoby DL, German P, Heitner SB, Kupfer S, Lutz JD, Malik FI, Meng L, Wohltman A, Abraham TP; SEQUOIA-HCM Investigators *. Dosing and Safety Profile of Aficamten in Symptomatic Obstructive Hypertrophic Cardiomyopathy: Results From SEQUOIA-HCM. J Am Heart Assoc. 2024 Aug 6;13(15):e035993. doi: 10.1161/JAHA.124.035993. Epub 2024 Jul 26. PMID 39056349
- [Derived] Maron MS, Masri A, Nassif ME, Barriales-Villa R, Arad M, Cardim N, Choudhury L, Claggett B, Coats CJ, Dungen HD, Garcia-Pavia P, Hagege AA, Januzzi JL, Lee MMY, Lewis GD, Ma CS, Michels M, Olivotto I, Oreziak A, Owens AT, Spertus JA, Solomon SD, Tfelt-Hansen J, van Sinttruije M, Veselka J, Watkins H, Jacoby DL, Heitner SB, Kupfer S, Malik FI, Meng L, Wohltman A, Abraham TP; SEQUOIA-HCM Investigators. Aficamten for Symptomatic Obstructive Hypertrophic Cardiomyopathy. N Engl J Med. 2024 May 30;390(20):1849-1861. doi: 10.1056/NEJMoa2401424. Epub 2024 May 13. PMID 38739079
- [Derived] Coats CJ, Maron MS, Abraham TP, Olivotto I, Lee MMY, Arad M, Cardim N, Ma CS, Choudhury L, Dungen HD, Garcia-Pavia P, Hagege AA, Lewis GD, Michels M, Oreziak A, Owens AT, Tfelt-Hansen J, Veselka J, Watkins HC, Heitner SB, Jacoby DL, Kupfer S, Malik FI, Meng L, Wohltman A, Masri A; SEQUOIA-HCM Investigators. Exercise Capacity in Patients With Obstructive Hypertrophic Cardiomyopathy: SEQUOIA-HCM Baseline Characteristics and Study Design. JACC Heart Fail. 2024 Jan;12(1):199-215. doi: 10.1016/j.jchf.2023.10.004. Epub 2023 Nov 29. PMID 38032573